CLINICAL TRIAL: NCT01579513
Title: Corticosteroid Therapy in Neonates Undergoing Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro16545; R01HL112968 (NIH)
Record Dates: First submitted 2012-04-13; First posted 2012-04-18 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Congenital Heart Disease; Disorder of Fetus or Newborn
Keywords: Cardiopulmonary Bypass (CPB); System Inflammatory Response; inflammation; Methylprednisolone; Neonates; Steroid; Cardiac Surgical Procedures; Children; Infants; Pediatrics; Glucocorticoid; Heart Disease; Heart Defects, Congenital; Cardiovascular Diseases; Cardiovascular Abnormalities; Corticosteroid; methylprednisolone Hemisuccinate; Hormones; Physiological Effects of Drugs; Randomized Clinical Trial
MeSH Terms: conditions — Heart Defects, Congenital; Fetal Diseases; Inflammation; Heart Diseases; Cardiovascular Diseases; Cardiovascular Abnormalities | interventions — Methylprednisolone; Adrenal Cortex Hormones; Steroids; Glucocorticoids; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraoperative Methylprednisone (Active Comparator): Neonates with congenital heart disease requiring surgery utilizing cardiopulmonary bypass(CPB) in the first month of life that receive one dose of intravenous methylprednisolone (30 mg/kg) during anesthetic induction.
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): Neonates with congenital heart disease requiring surgery utilizing cardiopulmonary bypass (CPB) in the first month of life that receive one dose of placebo (normal saline) during anesthetic induction.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone at a dose of 30 mg/kg body weight and a concentration of 62.5 mg/cc. The study drug will be delivered in a blinded fashion to the anesthesiologist and will be administered intravenously with the induction of anesthesia.
  Other Names: Solulmedrol; Medrol; Corticosteroid; Steroid; Glucocorticoid
  Arms: Intraoperative Methylprednisone
Drug: Placebo — Normal saline will be drawn up in an identical volume to that needed for active study drug. The study drug will be delivered in a blinded fashion to the anesthesiologist and will be administered intravenously with the induction of anesthesia.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Although cardiopulmonary bypass (heart-lung machine) is a necessary component of heart surgery, it is not without consequences. Cardiopulmonary bypass initiates a potent inflammatory response secondary to the body's recognition of the abnormal environment of the heart-lung machine. This inflammatory response may lead to poor heart, lung and kidney function after the heart surgery. This is turn can lead to longer times on the ventilator (breathing machine), the need for higher doses of heart medications, a longer stay in the intensive care unit and even death. This is particularly true in infants less than one month of age due to their size and the immaturity of their organs. The appreciation of the post-cardiopulmonary bypass inflammatory response has resulted in a number of interventions directed at its reduction. No therapy has been recognized as the standard of care; however steroid therapy has been applied most often despite unclear evidence of a benefit. This study aims to determine if steroids improve the outcomes of babies undergoing heart surgery.

DETAILED DESCRIPTION:
This study is a multi-institutional randomized double-blind placebo controlled trial of the use of glucocorticoids to improve the clinical course of neonates following cardiac surgery. Cardiopulmonary bypass (CPB) is critical to cardiac surgery, but the pathophysiologic processes engendered by CPB play an important role in post-operative recovery. The use, doses and schedule of glucocortiocoid administration to ameliorate these CPB induced processes is highly variable and without clear data to provide direction. The Primary Aim of this study is to compare the effects of intraoperative methylprednisolone to placebo on a composite morbidity-mortality outcome following neonatal CPB. Secondary Endpoints include: inotropic requirements, incidence of low cardiac output syndrome, fluid balance, ICU stay parameters, levels of inflammatory molecules, neuro-developmental outcomes, and safety parameters. The study will focus on neonates because their post-CPB clinical course is typically more severe, and that high level of severity itself provides a substrate for identifying the positive effects of a particular therapy. Finally, a therapy identified as beneficial has the greatest potential for benefit in this vulnerable population

ELIGIBILITY:
Inclusion Criteria:

* Age < 1 month
* Male and female patients who are scheduled to undergo cardiac surgery involving CPB

Exclusion Criteria:

* Prematurity: < 37 weeks post gestational age at time of surgery
* Treatment with intravenous steroids within the two days prior to scheduled surgery.
* Participation in research studies involving the evaluation of investigational drugs within 30 days of randomization.
* Suspected infection that would contraindicate steroid use (eg - Herpes)
* Known hypersensitivity to IVMP or one of its components or other contraindication to steroid therapy (eg - gastrointestinal bleeding).
* Preoperative use of mechanical circulatory support or active resuscitation at the time of proposed randomization.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2012-06; Primary Completion 2018-05-25 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Graham, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia
  - Medical University of South Carolina, Pediatric Cardiology, Charleston, South Carolina

REFERENCES:
- [Background] Graham EM, Atz AM, Butts RJ, Baker NL, Zyblewski SC, Deardorff RL, DeSantis SM, Reeves ST, Bradley SM, Spinale FG. Standardized preoperative corticosteroid treatment in neonates undergoing cardiac surgery: results from a randomized trial. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1523-9. doi: 10.1016/j.jtcvs.2011.04.019. Epub 2011 May 20. PMID 21600592
- [Background] Seghaye MC. The clinical implications of the systemic inflammatory reaction related to cardiac operations in children. Cardiol Young. 2003 Jun;13(3):228-39. doi: 10.1017/s1047951103000465. No abstract available. PMID 12903869
- [Background] Seghaye MC, Heyl W, Grabitz RG, Schumacher K, von Bernuth G, Rath W, Duchateau J. The production of pro- and anti-inflammatory cytokines in neonates assessed by stimulated whole cord blood culture and by plasma levels at birth. Biol Neonate. 1998;73(4):220-7. doi: 10.1159/000013980. PMID 9551188
- [Background] Checchia PA, Bronicki RA, Costello JM, Nelson DP. Steroid use before pediatric cardiac operations using cardiopulmonary bypass: an international survey of 36 centers. Pediatr Crit Care Med. 2005 Jul;6(4):441-4. doi: 10.1097/01.PCC.0000163678.20704.C5. PMID 15982431
- [Background] Robertson-Malt S, Afrane B, El Barbary M. Prophylactic steroids for pediatric open heart surgery. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD005550. doi: 10.1002/14651858.CD005550.pub2. PMID 17943866
- [Background] Pasquali SK, Hall M, Li JS, Peterson ED, Jaggers J, Lodge AJ, Marino BS, Goodman DM, Shah SS. Corticosteroids and outcome in children undergoing congenital heart surgery: analysis of the Pediatric Health Information Systems database. Circulation. 2010 Nov 23;122(21):2123-30. doi: 10.1161/CIRCULATIONAHA.110.948737. Epub 2010 Nov 8. PMID 21060075
- [Background] Pasquali SK, Li JS, He X, Jacobs ML, O'Brien SM, Hall M, Jaquiss RD, Welke KF, Peterson ED, Shah SS, Gaynor JW, Jacobs JP. Perioperative methylprednisolone and outcome in neonates undergoing heart surgery. Pediatrics. 2012 Feb;129(2):e385-91. doi: 10.1542/peds.2011-2034. Epub 2012 Jan 23. PMID 22271697
- [Background] Clarizia NA, Manlhiot C, Schwartz SM, Sivarajan VB, Maratta R, Holtby HM, Gruenwald CE, Caldarone CA, Van Arsdell GS, McCrindle BW. Improved outcomes associated with intraoperative steroid use in high-risk pediatric cardiac surgery. Ann Thorac Surg. 2011 Apr;91(4):1222-7. doi: 10.1016/j.athoracsur.2010.11.005. PMID 21440149
- [Derived] Everett AD, Buckley JP, Ellis G, Yang J, Graham D, Griffiths M, Bembea M, Graham EM. Association of Neurodevelopmental Outcomes With Environmental Exposure to Cyclohexanone During Neonatal Congenital Cardiac Operations: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 May 1;3(5):e204070. doi: 10.1001/jamanetworkopen.2020.4070. PMID 32374395

RESULTS

PARTICIPANT FLOW:
Period: Primary Hospitalization
Arm/Group | Intraoperative Methylprednisone | Placebo
Started | 91 | 99
Completed | 81 | 95
Not Completed | 10 | 4
Period: 1 Year Neurodevelopmental Follow up
Arm/Group | Intraoperative Methylprednisone | Placebo
Started | 81 | 95
Completed | 61 | 68
Not Completed | 20 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraoperative Methylprednisone | Placebo | Total
Number analyzed (Participants) | 81 | 95 | 176
Age, Continuous [Mean (Standard Deviation); unit: days] | 9.1 (5.4) | 8.2 (5.6) | 8.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 46 | 60 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 77 | 87 | 164
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 27 | 49
  White | 55 | 60 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 81 | 95 | 176
Weight at surgery [Mean (Standard Deviation); unit: Kg] — Weight in Kg at the time of surgery
  Kg | 3.2 (0.5) | 3.4 (0.5) | 3.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinically Derived Composite Morbidity-mortality Outcome
Description: The composite morbidity-mortality outcome will be met if any of the following occur after surgery but before hospital discharge: death, cardiac arrest, extracorporeal membrane oxygenation, renal insufficiency (creatinine more than two times normal), hepatic insufficiency (aspartate aminotransferase or alanine aminotransferase more than two times normal), or rising lactic acidosis (>5mmol/L). This outcome was choosen because death rarely occurs in this population. We have found this endpoint to be highly associated with other important clinical outcomes in this population.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Methylprednisone | Placebo
Number analyzed (Participants) | 81 | 95
Participants | 27 | 40

2. Secondary Outcome: Duration of Mechanical Ventilation Post Cardiac Surgery.
Description: Amount of time on mechanical ventilation following cardiac surgery
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intraoperative Methylprednisone | Placebo
Number analyzed (Participants) | 81 | 95
Days | 4 [3 to 7] | 5 [3 to 8]

3. Secondary Outcome: Intensive Care Unit Stay
Description: Amount of time in the intensive care unit following cardiac surgery
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Intraoperative Methylprednisone | Placebo
Number analyzed (Participants) | 81 | 95
Days | 11 [7 to 18] | 11 [7 to 20]

4. Secondary Outcome: Hospital Stay
Description: Total duration of hospital stay following cardiac surgery
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Intraoperative Methylprednisone | Placebo
Number analyzed (Participants) | 81 | 95
Days | 20 [13 to 35] | 22 [12 to 35]

5. Secondary Outcome: Neurodevelopmental Outcome
Description: Bayley Scales of Infant and Toddler Development version 3 at 1 year. Cognitive, language, and motor composite scores will be used. The general population has a mean of 100 with a standard deviation of 15 for each composite score. Higher scores are better. The minimum composite score is 46 and maximum 154.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intraoperative Methylprednisone | Placebo
Number analyzed (Participants) | 61 | 68
score on a scale
  Cognitive Domain | 105 (15) | 104 (14)
  Language Domain | 101 (15) | 100 (13)
  Motor Domain | 90 (16) | 91 (19)

ADVERSE EVENTS:
Time Frame: For the entirety of the initial neonatal hospitalization, an expected average of up to 5 weeks
Description: Death or the use of extracorporeal membrane oxygenation
Arm/Group | Intraoperative Methylprednisone | Placebo
All-Cause Mortality (participants affected / at risk) | 5/81 | 6/95
Serious Adverse Events (participants affected / at risk) | 4/81 | 11/95
Other Adverse Events (participants affected / at risk) | 2/81 | 2/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Methylprednisone (N=81) | Placebo (N=95)
Extracorporeal membrane oxygenation (Cardiac disorders) | 4 | 11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Methylprednisone (N=81) | Placebo (N=95)
Insulin therapy (Endocrine disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Nearly one third of the subjects received additional steroids in the early postoperative period, potentially diminishing the ability to detect both beneficial and adverse effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT01579513/Prot_SAP_000.pdf